CLINICAL TRIAL: NCT02208193
Title: Alzheimer's Disease and Healing Gardens: Study of the Cognitive and Psycho-behavioral Effects of an Artistic Dimension
Brief Title: Alzheimer's Disease, Art and Garden
Acronym: JAZ ART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-A00139-38
Record Dates: First submitted 2014-07-22; First posted 2014-08-04 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease Art Healing gardens Discourse analysis
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy controls group (Experimental): Healthy volunteers
  Interventions: Behavioral: Cognitive and psycho-behavioral effects of an artistic dimension
- Alzheimer subjects group (Experimental): Group A "Alzheimer group": patients with mild to severe stages of Alzheimer's disease: subgroup A1 "Alzheimer group hospitalized at the Paul Spillmann Centre (Centre Paul Spillmann, CPS)" (CHU de Nancy, France); subgroup A2 "Alzheimer group monitored at the Resource and Research Memory Centre (Centre Mémoire de Ressources et de Recherche, CMRR)" (CHU de Nancy, France)
  Interventions: Behavioral: Cognitive and psycho-behavioral effects of an artistic dimension

INTERVENTIONS:
Behavioral: Cognitive and psycho-behavioral effects of an artistic dimension

SUMMARY:
Gardens and art represent public spaces and support venues of interactions and emotions, seeking not only a variety of conversational themes but also various cognitive skills such as mnemonic skills. The cognitive and psycho-behavioral effects of art and the garden, jointly associated and made available to patients suffering from Alzheimer's disease, need to be evaluated.

MAIN OBJECTIVE Delineate the psychological scaffolding virtues of art and garden on cognitive and emotional processes by means of interview analyses in Alzheimer patients and control subjects based on the " art, memory and life " garden.

SECONDARY OBJECTIVES Adapt eco-psychosocial approaches of care management to Alzheimer patients:

* create assessment methods of:
* the therapeutic efficacy of the design of the " art, memory and life " garden,
* the perception of an artistic dimension in the living environment of those with Alzheimer's disease,
* establish:
* workshop applications using art and the garden for therapeutic purposes,
* general recommendations for the layout of the garden. PRIMARY ENDPOINT Quantitative data of discursive productions stemming from Interlocutory Logic (Trognon and Batt, 2007, 2010, 2011) for the analysis of interactive behaviors and the assessment of parameters including esthetic appraisals, well-being, mnemonic and emotional processes (frequency and nature of these processes) as well as spatio-temporal orientation.

SECONDARY ENDPOINTS

* Scores obtained in standard neuropsychological tests, in particular to assess spatio-temporal orientation (Folstein MMSE),
* Scores obtained with the " MemoArtZ " tool (MAZ) to evaluate the memorization of artistic elements of the garden,
* Scores from the " General Esthetic Preference " (GEP) tool to evaluate the consistency of general esthetic appreciations,
* Score obtained with the specific mood assessment scale (CSDD) for subjects in group A,
* Score obtained with the specific assessment of emotional events scale (AES) for all subjects.

RESEARCH METHODOLOGY

Open, monocentric, controlled (group of healthy control subjects) study.

Population: 2 groups:

Group A "Alzheimer group": patients with mild to severe stages of Alzheimer's disease: subgroup A1 "Alzheimer group hospitalized at the Paul Spillmann Centre (Centre Paul Spillmann, CPS)" (CHU de Nancy, France); subgroup A2 "Alzheimer group monitored at the Resource and Research Memory Centre (Centre Mémoire de Ressources et de Recherche, CMRR)" (CHU de Nancy, France) Group B "healthy control group": healthy volunteers

Therapeutic fallouts of this study will benefit Alzheimer patients in terms of better care management, notably: i) by determining the design, conception and layout of the gardens destined to these patients, ii) by developing the introduction of an artistic dimension to the design of such healing gardens and in their living environment, iii) by establishing workshop application perspectives using the contemplation of works of art and the garden for therapeutic purposes.

DETAILED DESCRIPTION:
RESEARCH METHODOLOGY / EXPERIMENTAL DESIGN

Open, monocentric, controlled (group of healthy control subjects) study.

Population: 2 groups:

Group A "Alzheimer group": patients with mild to severe stages of Alzheimer's disease: subgroup A1 "Alzheimer group hospitalized at the Paul Spillmann Centre (Centre Paul Spillmann, CPS)" (CHU de Nancy, France); subgroup A2 "Alzheimer group monitored at the Resource and Research Memory Centre (Centre Mémoire de Ressources et de Recherche, CMRR)" (CHU de Nancy, France) Group B "healthy control group": healthy volunteers

SPECIFIC ASSESSMENT PROCEDURES

TASKS SPECIFIC TO THE STUDY: MATERIALS

Interview methodology: The interrelationships between garden, art, cognition and behavior will be assessed. The endpoints of these dimensions will be achieved by an analysis of subject-psychologist interactions via interviews in the garden (in-context) and in out-of-context mnemonic interviews. These interviews will be recorded and transcribed verbatim. The interest of juxtaposing these two interview situations, in a comparative analysis of interactional production, is to be able to access different cognitive skills in order to analyze these skills. All of the data will be extracted through the quantitative analysis of discursive productions stemming from Interlocutory Logic (Trognon and Batt, 2007, 2010, 2011). The investigators analyses will consist, on the one hand, of exploring the public production of private thoughts of the subject (cognition and emotions) and secondly, to modelize interactive behaviors. The interlocutory space will be both referential and modal. All in all, the investigators will observe and analyze the eventual discursive productions of the subject in reference to the "art, memory and life" garden, whether they are related to the subject's experiences in the garden (in-context), to the narrative situation in recounting his or her experience in the garden (out-of-context) or to the spontaneous use of the garden for subjects in group A1. The implemented approach will have a strong ecological perspective.

Interlocutory logic is an analysis method developed in the INTERPSY laboratory . This pragmatic-dialogic method analyzes discourse in situations of interaction. This analytical process is aimed at expliciting the basic components of communication, interlocutory management and socio-cognitive-discursive events occurring in conversations.

For subjects in Group A:

Mood assessment: Cornell Scale for Depression in Dementia (CSDD, Cornell, 1988), translated into French.

For subjects in Group A and in Group B

* Assessment of emotional events: Apathy Scale: Marin's Apathy Evaluation Scale (AES)
* Questionnaire on artistic and cultural activities (ACA) pertaining to all artistic and cultural activities that the subject appreciates and/or is engaged in or has engaged in.
* Assessment of general esthetic preferences: "General Esthetic Preference" (GEP) tool
* Designed along the lines of those used by Kawabata and Zeki and by Halpern et al. for their respective studies (Kawabata and Zeki, 2010; Halpern et al., 2008).
* Materials: photographs representing works of art - paintings and sculptures - belonging to three styles: figurative, stylized or abstract, each representing categories - living or non-living.
* Task to be performed by the subject: for each photograph presented, the subject's task is to express an esthetic judgment using a visual analogue scale. After collecting the subject's esthetic judgment, his or her esthetic emotions will be assessed through two propositional questions.
* Objective: Document the feelings relative to the person's preference for a certain artistic style.

Interview-discovery and interview-knowledge of the garden (in-context) (30 min per interview): During the walk-through, the subject, accompanied by the psychologist, will observe the entire garden and its artistic elements. The subject will be queried through a discussion aimed at promoting the expressing of immediate reactions on the artistic dimensions. The analytical approach will enable to assess:

* the esthetic preferences of the artistic elements integrated in the garden
* the mnemonic and emotional processes (nature and frequency) that are mobilized during the contemplation of the elements of the garden, whether vegetation or artistic.
* the expressions of well-being and curiosity prompted by the works of art
* the mnemonic processes referring to temporality and space

Out-of-context assessments (90 min per assessment):

* Mnemonic interview (about 30 min): in a closed office blinded to the outside, the psychologist invites the subject to recall what he or she has experienced in the garden. In other words, the subject is asked to narrate an experience outside of its context. In this situation, the context must be formalized verbally which leads to the mobilization of cognitive skills other than those mobilized in the first in-context situation.
* General esthetic preferences (GEP tool): This assessment will reveal the perseverance for certain esthetic preferences or, conversely, the detachment relative to certain styles or categories addressed prior to the first walk in the garden.
* Mnemonic aspects of artistic elements " MémoArtZ " (MAZ) tool:
* Task to be performed by the subject: view photographs representing the various works of art discovered in the garden, inserted amidst distractive elements.
* Instructions: "Show me the photograph that represents an item you saw in the garden".
* Aim: the analysis will enable to objectify potential encoded memory recalls referring to the artistic elements of the garden.
* The mnemonic processes regarding temporality and space will also be brought to light through exchanges initiated by open questions, particularly around the theme of the current season of the year. The investigators will observe whether the fact of having been in the garden allows the subject to change and readjust his or her eventually inadequate response given at the MMSE (context aid).
* Mood assessment (CSDD) for subjects in group A only
* Assessment of emotional events (AES) for subjects in groups A and B.

ASSESSMENT SCHEDULE SPECIFIC TO THE RESEARCH

Group A " Alzheimer Group "

Subgroup A1 " Alzheimer group hospitalized at the Paul Spillmann Centre "

Inclusion visit With the investigator/physician

* Explanation of the objective and conduct of the research
* Upon participation consent: provision of the information document and of the consent form and signing of the latter
* Informing of the trusted person or primary caregiver (with provision of an information document)
* If patient consent: Informing of the attending physician
* Validation of inclusion and non-inclusion criteria

With the psychologist: T0:

* CSDD and AES scales
* ACA questionnaire
* GEP assessment

Visit 1 (as soon as possible after the inclusion visit)

Takes place in 2 stages on the same day:

* T1: Interview-discovery of the garden (in-context)
* T1+: Out-of-context assessment (mnemonic interview, GEP, MAZ, MMSE, CSDD, AES)

Spontaneous use of the garden

Visit 2 (after a three-day period of spontaneous use of the garden, consecutive or not, or from the 4th day onward within a maximum delay of 10 days after visit 1)

* T2: Interview-knowledge of the garden (in-context)
* T2+: out-of-context interview (mnemonic interview, GEP, MAZ, MMSE, CSDD, AES)

Subgroup A2 "Alzheimer group monitored at the Resource and Research Memory Centre (CMRR) "

At the CMRR with the investigator/physician:

* Verification of inclusion and non-inclusion criteria in light of medical records
* Upon participation consent: provision of the information document and the consent form
* Informing of the trusted person or primary caregiver (with provision of an information document)
* If patient consent: treating physician will be informed
* Scheduling of an appointment at the CPS

Visit 1 (over a single day, at the CPS)

Inclusion work-up with the investigator/physician of the CPS:

* Presentation of the study and careful reading of the information document
* Upon participation consent: signing of the consent form
* The person of trust or primary caregiver will be informed (an information document will be delivered)
* If patient consent: Informing of the attending physician
* Validation of inclusion and non-inclusion criteria

With the psychologist:

- T0: CSDD and AES scales ACA questionnaire GEP assessment

* T1: Interview-discovery of the garden (in-context)
* T1+: Out-of-context assessment (mnemonic interview, GEP, MAZ, MMSE, CSDD, AES)

Visit 2 (without use of the garden) within a maximum delay of 10 days after visit 1

* T2: Interview-knowledge of the garden (in-context)
* T2+: out-of-context interview (mnemonic interview, GEP, MAZ, MMSE, CSDD, AES)

Group B: " healthy control group "

Visit 1 (over a single day, at the CPS)

With the investigator/physician: inclusion work-up:

* Presentation of the study and careful reading of the information document
* Upon participation consent: signing of the consent form
* Validation of inclusion and non-inclusion criteria

With the psychologist:

-T0: Neuropsychological assessment (90 min): neuropsychological tests used in routine clinical practice CSDD and AES scale ACA questionnaire GEP assessment

* T1: Interview-discovery of the garden (in-context)
* T1+: out-of-context assessment (mnemonic interview, GEP, MAZ, MMSE, CSDD, AES)

Visit 2 (without use of the garden) within a maximum delay of 10 days after visit 1

* T2: Interview-knowledge of the garden (in-context)
* T2+: out-of-context interview (mnemonic interview, GEP, MAZ, MMSE, CSDD, AES) TOTAL NUMBER OF PARTICIPANTS Taking into account situations leading to permanent study discontinuations, 60 subjects will be included: 40 patients (group A) and 20 control subjects (group B)

DURATION OF THE STUDY Duration of inclusion period: 3 years Duration of participation: maximum 8 weeks for the patients (including the follow-up period); 11 days for control subjects Total duration time: 38 months (including analysis period and presentation of data)

STATISTICAL ANALYSIS The descriptive analysis will be performed by computing frequencies for categorical variables and mean and standard deviation or median and extreme values for continuous variables. The analysis will include a comparison of the different time periods of the study. Between-group comparison of frequencies (sick patients versus healthy subjects or paired series at different study times) will be performed by a Fisher Chi2 test or McNemar test, comparison of means by a nonparametric test or a paired t-test for paired series according to the conditions of application of the tests. The alpha risk is set at 5% for all analyses. An a posteriori power calculation will be performed retrospectively for all statistical tests. The analysis will be carried out using the SAS version V9.3 software package.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 to 100 years
* able to walk independently, that is to say without recourse to aid, whether human or technical, except for a simple cane
* have never been in the garden " art, memory and life " of the Paul Spillmann Centre
* gave their written consent after receiving clear and intelligible written and oral information
* with a diagnosis of a probable mild to severe stage of Alzheimer's disease according to NINCDS-ADRDA diagnostic criteria (McKhann et al., 1984) within the last 2 months prior to inclusion
* score less than or equal to 4 on the Hachinski Ischemic Scale (Hachinski et al., 1984) within the last 2 months prior to inclusion
* Folstein MMSE score between 7 and 24 inclusively within the last 2 months prior to inclusion
* score of 4, 5 or 6 on the Reisberg Global Deterioration Scale (Reisberg et al., 1982) within a 2-month delay prior to inclusion
* specific drug treatment for Alzheimer's disease, unchanged since at least 2 months (cholinesterase inhibitor and memantine)
* no change in psychotropic treatment within 48 hours prior to inclusion

Exclusion Criteria:

* lack of insurance coverage
* sensory deficit interfering with the designated tasks in the study
* phasic disorders interfering with the designated tasks in the study
* history of head trauma (with loss of consciousness)
* chronic alcoholism
* refusal or inability to obtain the informed written consent of the subject
* persons subject to a legal protection order
* severe depression: score > 20 on the GDS (Geriatric Depression Scale) scale at inclusion
* other neurological or psychiatric disorders potentially affecting the assessment
* current or planned participation to other research involving neuropsychological evaluations and/or drug trial, up until the end of the current study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-10 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Comparaison of the number of language acts in each category between AD and controls subjects | visit2 ( 10 days maximum after visit 1)
  Each interaction between a subject and the psychologist is distributed into a interlocutory analysis table (Trognon and Batt, 2010 ; Batt, Trognon, Rivasseau-Jonveaux, Vernant and Jonveaux, 2014) where each utterance is noticed by its speech turn and its speech act. The second consists of a force (for example, an assertive force, as when I was eight, I loved the garden my parents owned) and a propositional content (for example, a feeling in its episodic context). Propositional content will be described according to its stimulus (for example, a kind of flower growing in the garden, a sculpture put into some place, etc.), to the interaction where it is produced and, more crucially, to the level of memory (procedural/semantics/episodics) it involves. These are the variables that will be then compared in using usual statistics between paired AD and control subjects at visit 1 and 2

SECONDARY OUTCOMES:
Scores obtained in standard neuropsychological tests, in particular to assess spatio-temporal orientation (Folstein MMSE), | visit2 ( 10 days maximum after visit 1)
Scores obtained with the " MemoArtZ " tool (MAZ) to evaluate the memorization of artistic elements of the garden, | visit2 ( 10 days maximum after visit 1)
Scores from the " General Esthetic Preference " (GEP) tool to evaluate the consistency of general esthetic appreciations, | visit2 ( 10 days maximum after visit 1)
obtained with the specific mood assessment scale (CSDD) for subjects in group A | visit2 ( 10 days maximum after visit1)
Score obtained with the specific assessment of emotional events scale (AES) for all subjects. | visit2 ( 10 days maximum after visit 1)

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse Rivasseau Jonveaux, MD, Principal Investigator — CHU NANCY
Locations (1):
- CHU Nancy, Nancy, France